CLINICAL TRIAL: NCT04466527
Title: Laser Treatment for the Clinical Improvement of Acne Vulgaris: A Self-Controlled Trial
Brief Title: Laser Treatment of Moderate to Severe Acne Vulgaris
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Dieter Manstein, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P000838
Record Dates: First submitted 2020-07-02; First posted 2020-07-10 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Acne Vulgaris
Keywords: Acne; Acne Vulgaris; Laser; Cystic Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Subjects in this arm will undergo laser treatment on their active acne vulgaris lesions. Subjects will serve as their own control.
  Interventions: Device: Laser Intervention

INTERVENTIONS:
Device: Laser Intervention — Subjects with undergo laser exposure of their active acne vulgaris.

SUMMARY:
In this study, we are enrolling subjects with moderate to severe acne vulgaris and investigating the use of a commercially available laser in treating acne.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able and willing to provide written informed consent and comply with the requirements of the study protocol;
2. In good general health, based on answers provided during the screening visit;
3. Subject must be able to read and understand English;
4. Any gender and any Fitzpatrick skin type;
5. Ages 18 through 40;
6. Subjects must have moderate to severe nodular active facial acne vulgaris (PGA 3 or 4)
7. Willing to sun protect treated area for the duration of enrollment in the study and 1 year after treatment;
8. Subjects must be ineligible for or have declined standard of care treatments (e.g. oral isotretinoin therapy).

Exclusion Criteria:

1. Participation in another investigational drug or device clinical trial in the past 30 days;
2. Currently undergoing or wish to begin or continue topical treatments;
3. Are pregnant or lactating;
4. History of allergic reaction to topical anesthesia;
5. Subjects may not have undergone oral isotretinoin therapy within the past 12 months;
6. Currently take oral antibiotic or oral therapy for acne;
7. History of keloidal or hypertrophic scarring;
8. Laser treatment in past six months;
9. History of poor wound healing;
10. Clinically significant abnormal findings or conditions which might, in the opinion of the Investigator, interfere with study evaluations or pose a risk to subject safety during the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-05-20 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Changes in Physician's Global Assessment (PGA) of Acne Severity | Change in PGA score between baseline visit and post procedural visit
  The physician will score the acne vulgaris based on the Physician's Global Assessment (PGA) scale. A score of 0 indicates that residual hyperpigmentation and erythema may be present; a score of 1 indicates that there are a few scattered comedones and a few small papules; a score of 3 indicates that more than half of the face is involved, that there are many comedones, papules, and pustules, and that one nodule may be present; a score of 4 indicates that the entire face is involved, covered with comedones, numerous papules and pustules, and a few nodules and cysts. The change in PGA score will be recorded at each of the 4 study visits, for up to

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Manstein, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Clinical Unit for Research Trials & Outcomes in Skin, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No